CLINICAL TRIAL: NCT07238322
Title: An Assessment of the Efficacy of Floretyrosine F 18 ([18F]FET) Positron Emission Tomography (PET) for Characterization of Progressive or Recurrent Glioma From Treatment Related Changes
Brief Title: [18F]FET PET for Characterization of Progressive or Recurrent Glioma From Treatment Related Changes
Status: Enrolling by invitation | Type: Observational
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 18F-TLX101-005
Record Dates: First submitted 2025-10-01; First posted 2025-11-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Retrospective Study; Glioma; Brain Neoplasms
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Retrospective review of patients with histologically confirmed or suspected glioma (Grades 1-4) who underwent [18F]FET PET imaging as part of routine clinical care following completion of primary treatment (surgery, radiation, and/or chemotherapy), and who demonstrated radiographic suspicion of progression or recurrence on conventional imaging.
  Interventions: Diagnostic Test: 18F(FET)PET

INTERVENTIONS:
Diagnostic Test: 18F(FET)PET — Imaging as part of routine care

SUMMARY:
This study is designed to prospectively analyze [18F]FET PET image data obtained retrospectively in the routine clinical care of glioma patients. The study will analyse the data from participants with grade (1-4) glioma after primary treatment according to local clinical practice and with suspicion of progression/recurrence on magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Signed patient informed consent with secondary use of data permitted. Pediatric patients (<18 years of age) will provide assent along with parental/legal guardian /caregiver consent
2. Male or Female of any age at the time of [18F]FET PET imaging. While there is no age restriction, it is expected that enrollment of patients ≤ 3 years old will be rare due to the very low incidence of glioma in this age group.
3. Documented histologic diagnosis or clinical suspicion of glioma (Grades 1-4) based on local clinical assessment.
4. Underwent [18F]FET PET imaging as part of routine clinical care after completion of primary treatment (surgery, radiation therapy, and/or chemotherapy).
5. Evidence of radiographic suspicion of recurrence or progression on MRI at the time of [18F]FET PET imaging.
6. The adult patient, 18 years of age or older, has received nominal injected dose of 4 to 7 mCi (148 - 259 MBq ) of [18F]FET per imaging time point.
7. The pediatric patients, 0-17 years old, must have received a pediatric dose adjusted based upon the patient's body weight.

Exclusion Criteria:

Participants will be excluded if they did not meet any of the inclusion criteria or institutional requirements for participation.

1. Did not meet all inclusion criteria.
2. Did not undergo [18F]FET PET imaging as part of routine clinical care.
3. Imaging data or associated clinical information is incomplete, non-evaluable, or of insufficient quality for analysis.
4. Any institutional or regulatory requirement that precludes data sharing or inclusion in retrospective research studies.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are enrolled in the study will be included in the FAS.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 4 months
  The performance of [18F]FET PET in its ability to differentiate between benign treatment-related changes (TRC) and recurrent glioma (Grades 1-4) in comparison to a composite standard of truth (CSOT) will be evaluated and sensitivity and specificity evaluated.

CONTACTS AND LOCATIONS:
Locations (4):
- University of California, San Francisco, San Francisco, California, United States
- Germany (2):
  - University Hospital Essen, Essen
  - Universityhospital Tuebingen, Tübingen
- The University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No